CLINICAL TRIAL: NCT02182453
Title: A Phase I, Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (1 to 100 mg) of BI 10773 in Healthy Male Volunteers
Brief Title: Single Rising Oral Doses of BI 10773 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.5
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 10773 - single rising dose (Experimental)
  Interventions: Drug: BI 10773 - single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 10773 - single rising dose
  Arms: BI 10773 - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 10773 administered to healthy Japanese male subjects with single rising oral doses (1, 5, 10, 25, and 100 mg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers who meet the following criteria:

  * Without clinically remarkable findings or clinically evident complications based on their concurrent illness, past medical history, physical examination, vital signs (blood pressure, pulse rate, and body temperature), 12-lead ECG, and laboratory test results
  * Age ≥20 and Age ≤35 years
  * Body Mass Index (BMI) ≥18.0 and ≤25.0 kg/m2
  * Persons who are willing to participate in this trial and who give their written consent before study initiation in accordance with the Good Clinical Practice (GCP)

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, body temperature, and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to a drug or its excipients)
* Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug before administration of the investigational product or during the trial
* Use of any drugs within 10 days before administration of the investigational product or during the trial
* Participation in another trial with an investigational drug within four months before administration of the investigational product or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse
* Drug abuse
* Blood donation (100 mL or more) within four weeks before administration of the investigational product or during the trial
* Excessive physical activities within one week before administration of the investigational product or during the trial
* Basically, a patient with a laboratory value outside the reference range of the clinical site will be excluded form the study. However, if the principal investigator does not see any problem for the subject to enter the study based on the result of assessment of physical examination and other clinical examination, the subject will be able to participate in the study. In this regard, however, subjects who meet one of the following criteria will be excluded from the study:

  * FPG (Fasting plasma glucose) ≥110mg/dL
  * eGFR (estimated glomerular filtration rate) <60
  * abnormal value of urinalysis
* Inability to comply with dietary regimen of the study centre
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for TdP (torsade de pointes) (e.g., heart failure, hypokalemia, family history of long QT syndrome)Samsung2014
* Renal glucosuria or elevated urinary glucose levels at screening (>15 mg/dl)
* Any abnormal finding in Kidney or patients who have history of renal disease
* Any other clinical conditions that investigator or sub-investigator judges that the subject is ineligible for study participation

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 7 days
Number of patients with abnormal changes in laboratory parameters | Baseline, day 2-4 and day 7
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate, and body temperature) | Baseline, day 1-4 and day 7
Number of patients with clinical significant changes in 12-lead ECG (electrocardiogram) | Baseline, day 1-4 and day 7
Assessment of tolerability on a 4-point scale | Day 4

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
tmax (time from dosing to maximum concentration) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
λz (terminal rate constant in plasma) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
t1/2 (terminal half-life of the analyte in plasma) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
MRTpo (mean residence time of the analyte in the body after po administration) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
CL/F (total clearance of the analyte in the plasma after extravascular administration) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Before and 10, 20, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 34, 48 72 hours after administration of study drug
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | 2 hours before and 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-34, 34-48, and 48-72 hours after administration of study drug
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | 2 hours before and 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-34, 34-48, and 48-72 hours after administration of study drug
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | 2 hours before and 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-34, 34-48, and 48-72 hours after administration of study drug